CLINICAL TRIAL: NCT05616429
Title: Alcat Based Elimination Diet for the Treatment of Irritable Bowel Syndrome; a Randomized Double Blind Sham Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Cell science systems (Unknown)
Responsible Party: Principal Investigator, Dr. Tal Engel, Principal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6834-20-TA-CTIL
Record Dates: First submitted 2022-10-26; First posted 2022-11-15 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Double blind randomized clinical trial (RCT) comparing Alcat based personal diet for the treatment of IBS versus "sham" standard balanced diet
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcat based personal diet (Experimental)
  Interventions: Dietary Supplement: Alcat based personal diet; Other: usual care
- Standard balanced diet (Sham Comparator)
  Interventions: Dietary Supplement: Standard balanced diet; Other: usual care

INTERVENTIONS:
Dietary Supplement: Alcat based personal diet — Alcat based personalized diet with dietician supervision and follow-up + usual care
  Arms: Alcat based personal diet
Dietary Supplement: Standard balanced diet — "Sham" standard balanced diet with dietician supervision and follow up + usual care.
  Arms: Standard balanced diet
Other: usual care — usual care

SUMMARY:
Irritable bowel syndrome (IBS) is the most common GI condition with global prevalence ranging between 10-20%. Although the exact cause is not known there are increasing insights concerning the possible multifactorial etiology including low grade inflammation, neuromodulation, dysbiosis, impaired integrity of the intestinal barrier and more.

Currently, it is believed that changes in the microbiota may activate mucosal innate immune responses, resulting in increased epithelial permeability, activated nociceptive sensory pathways, and dysregulation of the enteric nervous system.

Nearly two thirds of patients with IBS perceive their GI symptoms to be food related, hence, food intolerance may be important factor in the pathogenesis. Diet is a part of IBS treatment but adherence, on the one hand, and restriction, on the other, remain a major problem. [Chey WD, Am J Gastroenterol,2016].

Confocal laser endomicroscopy (CLE) is a technique that permits real-time detection and quantification of changes in intestinal tissues and cells, including increases in intraepithelial lymphocytes and fluid extravasation through epithelial leaks.

Based on CLE analysis of IBS patients with a suspected food intolerance, exposure to candidate food antigens caused immediate breaks, increased intervillous spaces, and increased IELs in the intestinal mucosa. These changes are associated with patient responses to exclusion diets. [Fritscher-Ravens A et al, Gastroenterology. 2019, Gastroenterology. 2014] This technic, also efficient according to former studies, is costly and invasive.

The Alcat Test is a lab based immune stimulation test in which a patient's WBC's (white blood cell) are challenged with various substances including foods, additives, colorings, chemicals, medicinal herbs, functional foods, molds and pharmaceutical compounds. The Alcat Test objectively classifies a patient's response to each test substance as reactive, borderline or non-reactive. Based on these classifications, a customized elimination/rotation diet may be designed.

DETAILED DESCRIPTION:
Diet therapies for IBS are becoming an important part of the treatment for patients with IBS [Lenhart A et al, J Neurogastroenterology Motil 2018] There are many types of elimination diets utilized by patients with IBS including personalized diets based upon mediator release testing and IgG (immunoglobulin G) antibody. These diets have the potential for tailor made personal diet but currently have little or no clinical evidence for efficacy.

Diet therapies, like medical therapies for IBS, should be properly evaluated in appropriate designed clinical trials.

It is also important to protect our patients with IBS from potentially ineffective, costly and unsafe intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Only adults (>18 years of age) meeting the Rome 4 Criteria for IBS D/M/U and who are willing to adhere to diet restrictions, will be eligible for entry into the study.
2. Patients with 'warning symptoms' (e.g., unexplained weight loss, history of GI cancer or inflammatory bowel disease, rectal bleeding etc) will be required to have had a detailed workup to exclude organic pathology prior to enrollment.
3. Participants will be allowed to continue their IBS medications (e.g., fiber, anti-spasmodics, antidepressants, loperamide, etc.) as long as they had been on stable doses for at least 30 days prior to entering the study and agreed not to change medications or dosages during the trial.
4. In addition, patients will be required to have active symptoms at the entry of the study as defined by having an IBSSSS score of >150 (0-500 scale).

Exclusion Criteria:

1. Patients will be excluded if they fulfill ROME 4 IBS C criteria
2. Have an inflammatory bowel disease, celiac or other inflammatory or gut disorder other than IBS.
3. Have active malignancy of any kind
4. If they are not able to eat PO
5. If they are Using NSAIDS more than once per month and within the 4 weeks prior to inclusion
6. If C reactive protein is above 2 times the normal value or if stool Calprotectin is above 200mcg/gr
7. If they had recent antibiotic use (within 1 month). -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome (IBS) Symptom Severity Scale questionnaire | 8 weeks
  decrease of 50 points. Values range: 0-500

SECONDARY OUTCOMES:
Irritable Bowel Syndrome Global Symptom Assessment (IBS-GSA) questionnaire | 4 and 8 weeks
  Compared to how you felt then, how would you rate your overall IBS symptoms during the past week? Possible answers are one of the following: Significantly relieved (+3); Moderately relieved (+2); A little bit relieved (+1); Unchanged (0); A little bit worse (-1); Moderately worse (-2); Significantly worse (-3).
  [ Rome Foundation]
Abnormal laboratory value - bio marker | 8 weeks
  decrease level - CRP (C reactive protein) milligrams per liter (mg/L)
Monitoring serum level of Syndecan-1 (Sdc1) ng/mL | 8 weeks
  Syndecan-1 (Sdc-1) is a type 1 transmembrane heparan sulfate proteoglycans that are implicated in maintenance of intestinal epithelial barrier. Sdc-1 is predominantly expressed by plasma cells and mucosal epithelial cells, such as intestinal epithelial cells.
  Changes of Sdc1 level in sera will be assessed primarily to the diet intervention and at the end of the diet after 8 weeks
Irritable Bowel Syndrome (IBS) Adequate Relief questionnaire | up to 8 weeks
  IBS-Adequate Relief (IBS-AR) is a dichotomous single item that asks participants "Over the past week have you had adequate relief of your IBS symptoms?
Irritable Bowel Syndrome Quality of life questionnaire - specific for IBS (IBS-QoL) | 8 weeks
  Changes from baseline to Week 8 in IBS-QOL total and subscale scores . Values: 34-170
Irritable Bowel Syndrome Global Improvement Scale (IBS-GIS) | up to 8 weeks
  Compared to the way you felt before you entered the study, have your IBS symptoms over the past 7 days been: 1) Substantially Worse, 2) Moderately Worse, 3)Slightly Worse, 4) No Change, 5) Slightly Improved, 6) Moderately Improved or 7) Substantially Improved. A responder is defined as a patient who answered "moderately improved" or "substantially improved".

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No